CLINICAL TRIAL: NCT06815601
Title: Neuromodulation After Spinal Cord Injury to Improve Limb Function
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Hang Jin Jo, Assistant Professor, State University of New York at Buffalo
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 00007259
Record Dates: First submitted 2025-01-24; First posted 2025-02-07 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-02

CONDITIONS: Spinal Cord Injury; Spinal Cord Injury Cervical
Keywords: spinal cord injury; SCI; Stimulation; Paralysis; rTMS; transcranial magnetic stimulation
MeSH Terms: conditions — Spinal Cord Injuries; Paralysis | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- rTMS (Active Comparator): rTMS will be administered and functional and physiological outcomes will be measured before and after each intervention.
  Interventions: Other: rTMS
- Sham rTMS (Sham Comparator): Sham rTMS will be administered and functional and physiological outcomes will be measured before and after each intervention.
  Interventions: Other: Sham rTMS
- rTMS with motor training (Active Comparator): Subjects will receive the rTMS with motor training for long-term up to 50 sessions. Motor training involves hand motor training.
  Interventions: Other: rTMS; Behavioral: Motor training

INTERVENTIONS:
Other: rTMS — Intermittent theta burst stimulation (iTBS) will be utilized since they have been reported to have a cortical neuromodulatory effect. The iTBS protocol will be applied over primary motor cortex to investigate its effect on corticospinal excitability and functional outcome. Theta burst stimulation (TBS) consists of bursts of pulses containing 3 pulses at 50 Hz (3 pulses per second) repeated at 200 ms intervals (5 Hz). During iTBS, a 2 second train of TBS is repeated every 10 seconds (600 pulses in 190 seconds).
  Other Names: iTBS
  Arms: rTMS; rTMS with motor training
Other: Sham rTMS — Sham iTBS protocols will be applied with the same parameters as in iTBS protocol. However, sham coil will be used.
  Other Names: Sham iTBS; Sham stimulation
  Arms: Sham rTMS
Behavioral: Motor training — The motor training will be focused on participant's hand motor function such as grasping function.
  Other Names: Exercise training; Hand training
  Arms: rTMS with motor training

SUMMARY:
The University at Buffalo (UB) Department of Rehabilitation Sciences is looking for adult volunteers with and without spinal cord injuries for a study on hand movement. The goal of the study is to learn about how the brain, nerves, and muscles of the body are connected and perform everyday tasks. This may help us to develop ways to improve the hand functions of people with spinal cord injuries.

DETAILED DESCRIPTION:
The main goal of rehabilitation strategies in humans with spinal cord injury (SCI) is to strengthen transmission in spared neural networks to restore functional movements. Recent evidence showed that neuromodulation approaches may increase the transmission in corticospinal pathway in humans with SCI and improve functional outcomes. Therefore, the investigators aim to investigate how the noninvasive brain stimulation protocols affects neuroplasticity of corticospinal pathway. Specifically, the investigators will use the repetitive transcranial magnetic stimulation (rTMS) to explore its effect. The investigators will investigate the effect of short-term and long-term rTMS application in individuals with SCI.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults between the ages of 18-75 years old who are right-handed
* Adults between the ages of 18-75 years old who have had a spinal cord injury (SCI)

Exclusion Criteria:

For both healthy individuals and those with SCI:

* Uncontrolled medical problems including pulmonary, cardiovascular or orthopedic disease
* Any debilitating disease prior to the SCI that caused exercise intolerance
* Ongoing major depression or altered cognitive status
* Metal plate in skull
* History of seizures
* Receiving drugs acting primarily on the central nervous system, which lower the seizure threshold such as antipsychotic drugs
* Pregnant females

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Motor evoked potentials (MEP) | For "rTMS" and "Sham rTMS", the time frame will be one day, before and after each session. For "rTMS with motor training", the time frame will be weekly up to 20 weeks.
  Transcranial magnetic stimuli (TMS) will be delivered through a figure-of-eight coil over primary motor cortex to the optimal scalp position for activation of hand muscles. The optimal scalp position will be determined by moving the coil in small steps along the hand representations of the primary motor cortex to find the region where the largest MEP can be evoked with the minimum intensity in the targeted muscle. Twenty MEPs will be collected and the peak-to-peak amplitude of MEP will be averaged across trials.

SECONDARY OUTCOMES:
Maximum voluntary contraction (MVC) | For "rTMS" and "Sham rTMS", the time frame will be one day, before and after each session. For "rTMS with motor training", the time frame will be weekly up to 20 weeks.
  Individuals will perform a MVC of the targeted hand muscle (first dorsal interosseous) through surface EMG electrodes. The investigators will collect two MVC trials and use the average of the two.
Power Grip Forces | For "rTMS" and "Sham rTMS", the time frame will be one day, before and after each session. For "rTMS with motor training", the time frame will be weekly up to 20 weeks.
  Power grip force will be measured with hand-held dynamometer.

CONTACTS AND LOCATIONS:
Overall Officials: Hang Jin Jo, PhD, Principal Investigator — State University of New York at Buffalo
Locations (1):
- The Kimball Tower at The State University of New York at Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No